CLINICAL TRIAL: NCT02046772
Title: Assessment of the Analgesic Efficacy of Morphine Chloride in Addition to a Low Dose Solution of Spinal Anaesthetic in Hemorrhoidectomy Compared to a Standard Dose of Spinal Local Anaesthetic. Simple Blind, Randomized, With Blinded Evaluation by Third Parties Clinical Trial.
Brief Title: Safety and Efficacy of the Addition of Morphine Chloride to a Low Dose of Bupivacaine as Intradural Anaesthetic for the Removal Surgery of the Hemorrhoids
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion para la Investigacion Biomedica del Hospital Universitario Principe de Asturias (Other)
Collaborators: Spanish Agency of Medicines and Health Products (Other Government); Spanish Health Ministry (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HUPA-EC-01-2012; 2012-000110-11 (EudraCT Number)
Record Dates: First submitted 2014-01-22; First posted 2014-01-28 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2014-08

CONDITIONS: Surgical Remove of Hemorrhoids
Keywords: hemorrhoidectomy; analgesia; anaesthetic; bupivacaine; morphine chloride
MeSH Terms: conditions — Agnosia | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Bupivacaine + Morphine Chloride (Experimental): People in this arm will receive treatment with morphine chloride in addition to a low dose solution of the local intradural anaesthetic bupivacaine.
  Interventions: Drug: Bupivacaine low dose; Drug: Morphine Chloride
- Bupivacaine standard dose (Active Comparator): People in this arm will receive treatment with the standard dose of the local intradural anaesthetic bupivacaine
  Interventions: Drug: Bupivacaine standard dose

INTERVENTIONS:
Drug: Bupivacaine low dose — A dose of morphine chloride added to a low dose solution of bupivacaine administered intradural
  Arms: Bupivacaine + Morphine Chloride
Drug: Bupivacaine standard dose — Single intradural standard dose of bupivacaine
  Arms: Bupivacaine standard dose
Drug: Morphine Chloride — A dose of morphine chloride added to a low dose solution of bupivacaine administered intradural
  Arms: Bupivacaine + Morphine Chloride

SUMMARY:
A single blind, randomized, with blinded evaluation by third parties clinical trial is carried out to assess the analgesic efficay of the addition of morphine chloride to a low dose solution of spinal local anaesthetic compared to a standard dose spinal anaesthetic in the haemorrhoid surgery.

The objective of this clinical trial is to assess if the experimental treatment is as efficacy as the standard treatment in the anesthetic and analgesic effects with less side effects, greater and earlier mobility after surgery and shortened the hospitalization.

DETAILED DESCRIPTION:
DESIGN OF THE TRIAL:

A multicentre, randomized, single-blind, with masked evaluationby third parties clinical trial.

The Clinical Pharmacology Unit will perform a permuted blocks randomization scheme for each of the two hospitals participating in the trial. The result of this randomization will be kept in this unit and will not be accessible to investigators. Investigators will receive a series of opaque sealed envelopes with a number corresponding to the order of entry of the patients into the trial. When the patient is in the operating room, investigators must open the envelope which contains the group of treatment assigned to that patient. The patient will not know in which intervention group is included. Investigator who performs the spinal puncture and investigator who collects the data and performs the evaluation will no be the same person. This will allow a blind evaluation.

OBJECTIVES:

Main objective:

To evaluate whether the addition of morphine chloride to a low dose solution of local intradural anaesthetic in patients undergoing hemorrhoids surgery produces an anaesthetic efficacy comparable to that produced by a standard dose of local intradural anaesthetic and an improvement of postoperative analgesic efficacy.

Secondary objectives:

* Earlier mobilization of the patient.
* Minor adverse effects.
* A shorter hospital stay of the patient.

TREATMENTS:

Two groups of treatment will be formed, experimental and comparator. The experimental group will receive 3mg of Bupivacaine with addition of 50 micrograms of Morphine Chloride.

The comparator group will receive 5 mg of Bupivacaine.

RESCUE TREATMENTS

If necessary before surgery, midazolam will be administered from 0.02 to 0.05 mg / kg intravenous (IV) depending on clinical response and after the patient is set in the surgical position, if necessary, an intravenous infusion of propofol will be administered at 0.5 - 2mg / kg / h. Sedative drugs with analgesic effects as opioids, ketamine, etc, will be avoided to not interfere with the main analgesic study assessment.

After surgery and during the hospitalization stay the rescue analgesia treatment will be administered only on demand. The rescue treatment allowed by protocol will be an intravenous administration of dexketoprofen up to 50 mg / 8 h and if insufficient, a rescue of 3 mg of morphine chloride will be administered. If morphine chloride is received, these patients will be recorded in the case report forms as inefficacy of the treatment. At home, after discharge, patients will receive rescue analgesia with capsules of dexketoprofen 25 mg / 8 h. (up to 75 mg a day).

SAMPLE SIZE:

66 patients ( 33 patients in the experimental group and 33 patients in the control group)

EFFICACY ASSESSMENT

Pain will be assessed using a visual analog scale (VAS from 0 to 10) at the beginning and end of surgery, at the arrival of resuscitation unit, after 10 and 30 minutes after arrival, during hospitalization stay out of the resuscitation unit and daily at home after discharge.

Doses required of rescue analgesia and hospitalization time will be recorded.

SAFETY ASSESSMENT

Basic monitoring as usual will be perfomed in the surgery room. Motor blockage will be assessed using the modified Bromage scale as follows: 1 = complete motor blocking, 2 = able to move feet only, 3 = patient move the feet and bend the knee, 4 = straight leg raises <30 ° or > 30 ° but not against resistance, 5 = lifts leg> 30 ° against resistance. This measure will be made after surgery in the surgery room and at the arrival and at one hour after resuscitation unit admission.

All the Adverse events will be reported.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hemorrhoidectomy.
* Age between 18 and 64.
* Both gender
* ASA I to III.
* With indication for spinal block.
* People capable to grant the informed consent.

Exclusion Criteria:

* Patients with allergies to the study drugs.
* Patients with any contraindication for performing a spinal technique (coagulation disorders, fever, intracraneal hypertension, abscess in the puncture site, etc..).
* Patients with previous neurological disorders.
* Pregnant women.
* Women who may be pregnant and do not have a negative pregnancy test.
* Breastfeeding women.
* Patients with uncapable to give informed consent.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2012-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Ruiz Castro, MD, PhD, Principal Investigator — Hospital Universitario Principe de Asturias
Locations (2):
- Spain (2):
  - Hospital Universitario Principe de Asturias, Alcalá de Henares, Madrid
  - Hospital del Henares, Coslada, Madrid

RESULTS

PARTICIPANT FLOW:
Groups:
- Bupivacaine + Morphine Chloride: People in this arm will receive treatment with morphine chloride (50 mcgr) in addition to a low dose solution of the local intradural anaesthetic bupivacaine (3mg).
  Bupivacaine low dose: A dose of morphine chloride added to a low dose solution of bupivacaine administered intradural.
  Morphine Chloride: A dose of morphine chloride added to a low dose solution of bupivacaine administered intradural.
- Bupivacaine Standard Dose: People in this arm will receive treatment with the standard dose of the local intradural anaesthetic bupivacaine (5mg).
  Bupivacaine standard dose: Single intradural standard dose of bupivacaine.
Period: Overall Study
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose
Started | 30 | 33
Completed | 30 | 33
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose | Total
Number analyzed (Participants) | 30 | 33 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.8 (10.5) | 51.3 (10.8) | 48.7 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 26
  Male | 17 | 20 | 37
Region of Enrollment [Number; unit: participants]
  Spain | 30 | 33 | 63
BMI [Mean (Standard Deviation); unit: Kg*m^-2] | 25.1 (3.3) | 27.2 (4) | 26.2 (3.9)
ASA [Number; unit: participants] — ASA is the clasification system created by the American Society of Anesthesiologists to set the risk of a patient that is about to receive surgery.
  The score range goes from I, where the patient is completely healthy, to VI, where the patient is extremely in life threatening.
  participants
    ASA I | 7 | 8 | 15
    ASA II | 22 | 25 | 47
    ASA III | 1 | 0 | 1
Number of haemorrhoidal packs removed [Number; unit: participants]
  1 haemorrhoidal pack | 8 | 12 | 20
  2 haemorrhoidal packs | 12 | 13 | 25
  3 haemorrhoidal packs | 8 | 8 | 16
  Unavailable | 2 | 0 | 2
Need of pre-surgery sedation [Number; unit: participants]
  Yes | 23 | 23 | 46
  No | 7 | 10 | 17
Duration of surgery [Mean (Standard Deviation); unit: minutes] | 28 (11.1) | 20.4 (9.2) | 24 (10.8)

OUTCOME MEASURES:

1. Primary Outcome: Measurement of Time to Start the Anaesthetic Effect
Description: To compare whether the addition of morphine chloride to a low dose intradural solution of the local anaesthetic bupivacaine is as effective as an administration of a single dose of bupivacaine.
Time Frame: First 20 minutes between administration and beginning of surgery
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose
Number analyzed (Participants) | 30 | 33
minutes
  Time to sensitive blocking | 2.1 (1.8) | 1.6 (1.5)
  Time to motor blocking | 7.7 (5.9) | 4.7 (3.3)

2. Primary Outcome: Measurement of the Analgesic Effect After Surgery by VAS From 0 to 10, Where 0 is no Pain and 10 is the Worst Pain Imaginable.
Description: To compare whether the addition of morphine chloride to a low dose solution of bupivacaine and improves the analgesic treatment than a single administration of bupivacaine.
Time Frame: Up to 72 hours from the end of the surgery in the hospital stay and during the next 7 days at home, after discharge
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose
Number analyzed (Participants) | 30 | 33
units on a scale
  VAS at the enter in the reanimation unit | 0.03 (0.1) | 0.15 (0.7)
  VAS after 10 minutes in reanimation unit | 0 (0) | 0.3 (1)
  VAS after 30 minutes in reanimation unit | 0.06 (0.3) | 0.72 (1.5)
  VAS day 1 after surgery | 1.5 (1.2) | 3.3 (2.2)
  VAS day 2 after surgery | 3.8 (2.8) | 4 (2.5)
  VAS day 3 after surgery | 3.7 (2.7) | 4.5 (2.3)
  VAS day 4 after surgery | 3.6 (2.6) | 4.4 (2.3)
  VAS day 5 after surgery | 3.6 (2.3) | 4 (2.2)
  VAS day 6 after surgery | 3.2 (2.6) | 3.5 (2.3)
  VAS day 7 after surgery | 2.5 (2.3) | 3 (2.2)

3. Secondary Outcome: Greater and Earlier Mobilization Measured by Bromage Scale.
Description: To assess whether the administration of morphine chloride in addition to a low dose solution of local intradural anaesthetic (bupivacaine) improves the mobilization of the patients after surgery more than the single intradural administration of bupivacaine.
  Total Score in the Bromage Scale goes from 1 to 5, where:
  1: complete motor blocking - 2: capable to move the feet - 3: moves the feet and bends the knee - 4: raise the leg straight more or less than 30 degrees but no against resistance - 5: raise the leg straight more than 30 degrees against resistance (no motor blocking)
Time Frame: During the first 24 hours after surgery and at the entry and exit of the resuscitation unit
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose
Number analyzed (Participants) | 30 | 33
units on a scale
  Bromage at the exit of surgery | 4 (1.3) | 3.7 (1)
  Bromage at the enter in the reanimation unit | 4.1 (1.1) | 3.8 (1)
  Bromage at the exit of the reanimation unit | 4.7 (0.4) | 4.8 (0.3)

4. Secondary Outcome: Number of Adverse Events
Description: To assess if the experimental treatment causes less, equal or more adverse events than the comparator treatment.
Time Frame: Up to 72 hours from the intervention and the hopitalary stay and during the next 7 days after discharge
Measure: Number; unit: participants
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose
Number analyzed (Participants) | 30 | 33
participants
  Pruritus | 2 | 0
  Urinary retention | 7 | 3
  Nausea/Vomits | 0 | 1
  Fever | 1 | 0

5. Secondary Outcome: Time of Hospitalization
Description: To see if the hospitalization time is shortened or not by the experimental treatment.
Time Frame: Up to 72 hours after the intervention
Measure: Number; unit: participants
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose
Number analyzed (Participants) | 30 | 33
participants
  1 day of hospitalization | 26 | 30
  2 days of hospitalization | 3 | 2
  3 days of hospitalization | 1 | 1

ADVERSE EVENTS:
Arm/Group | Bupivacaine + Morphine Chloride | Bupivacaine Standard Dose
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/33
Other Adverse Events (participants affected / at risk) | 10/30 | 4/33
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bupivacaine + Morphine Chloride (N=30) | Bupivacaine Standard Dose (N=33)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Urinary retention (Renal and urinary disorders) | 7 (7) | 3 (3)
Nausea or Vomits (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No